CLINICAL TRIAL: NCT05767307
Title: Danish Prostate Cancer Consortium Study-1 (DPCC-1): Multicenter Development of Liquid Biopsy Biomarkers for Early Detection of Prostate Cancer.
Brief Title: Danish Prostate Cancer Consortium Study-1
Acronym: DPCC-1
Status: Recruiting | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other); Odense University Hospital (Other); Herlev and Gentofte Hospital (Other)
Responsible Party: Sponsor
Organization: University of Aarhus (Other)
Other Study IDs: 1-10-72-85-22
Record Dates: First submitted 2023-02-08; First posted 2023-03-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (plasma, serum, and buffy coat) and urine (supernatant and pellet)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI-first: Biopsy naïve men referred to "MRI-first" due to suspicion of PC (elevated PSA and/or suspect DRE) at one of the following three major urology/uroradiology centers in Denmark: Aarhus University Hospital (AUH), Herlev & Gentofte Hospital (HH), and Odense University Hospital (OUH), where MRI and targeted biopsy is already implemented in clinical use.

SUMMARY:
The purpose of the study is to investigate if a new promising microRNA-based urine biomarker test for prostate cancer, called uCaP, is better than the current standard test (PSA) to identify men who would benefit from an MRI scan of the prostate. The study will include 2,500 men referred to MRI of the prostate at three major hospital centers in Denmark (Aarhus, Odense, and Herlev) and compare the accuracy of uCaP to PSA. Based on preliminary data it is expected that uCaP will be >20% better than PSA at identifying treatment-requiring cancer. Hence, uCaP could help to better pre-select men for MRI and thereby reduce unnecessary MRI scans, unnecessary prostate biopsies, as well as overdiagnosis and overtreatment of indolent PCs, while maintaining high sensitivity for aggressive PC that needs early detection and early treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Understand oral and written Danish.
* Referred to MRI (multi or bi-parametric) due to suspicion of PC at AUH, OUH, or HGH.

Exclusion Criteria:

* Previously diagnosed with PC or other urogenital cancers.
* Has one or more contraindications for MRI.
* Have had gender reassignment treatment.
* Blood PSA levels > 20 μg/l.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males referred to "MRI-first" due to suspicion of PC (elevated PSA and/or suspect DRE) at one of the following three major urology/uroradiology centers in Denmark: Aarhus University Hospital (AUH), Herlev & Gentofte Hospital (HGH), and Odense University Hospital (OUH).
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2040-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of MRI scans used to detect clinically significant PCs. | At recruitment completion, at year 3 in 2025
  Compare the total number of MRI scans required to detect clinically significant PC in the study population for the uCaP score vs. PSA or a combination of uCaP+PSA vs. PSA alone.
Clinically significant PC diagnoses compared to benign biopsies. | At recruitment completion, at year 3 in 2025
  Compare the number of patients diagnosed with clinically significant PC compared to the number of patients with benign biopsies (no cancer; i.e. unnecessary biopsy) for the uCaP score vs. PSA or a combination of uCaP+PSA vs. PSA alone.
Clinically significant PC diagnoses compared to clinically insignificant PC diagnoses. | At recruitment completion, at year 3 in 2025
  Compare the number of men diagnosed with clinically significant PC with the number of men diagnosed with clinically insignificant PC (i.e. overdiagnosed) for the uCaP score vs. PSA or a combination of uCaP+PSA vs. PSA alone.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus N, Aarhus
  - Herlev & Gentofte University Hospital, Hellerup
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fredsoe J, Glud E, Boesen L, Logager V, Poulsen MH, Pedersen BG, Borre M, Sorensen KD. Danish Prostate Cancer Consortium Study 1 (DPCC-1) protocol: Multicentre prospective validation of the urine-based three-microRNA biomarker model uCaP. BMJ Open. 2023 Nov 8;13(11):e077020. doi: 10.1136/bmjopen-2023-077020. PMID 37940151